CLINICAL TRIAL: NCT05396846
Title: MyGI Diet for Colorectal Cancer Prevention
Brief Title: My Best GI Eating Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Zora Djuric, Research Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HUM00197337; R01CA255743 (NIH)
Record Dates: First submitted 2022-05-19; First posted 2022-05-31 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Neoplasms
Keywords: Prevention; Diet
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be stratified by self-reported gender (male/female) and randomized across three study arms in a mixed block size, after baseline assessments are completed. Indeterminate gender will be classified as male for the purpose of randomization. The lists will be generated by the study statistician and opaque envelopes will contain the diet arm assignment for sequential participant IDs in the two strata.
Who Masked: Outcomes Assessor
Masking Description: All data and samples will be identified by a participant ID number and visit number. Results will be unblinded with regard to study arm assignment during statistical analysis only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eating Plan 1 (Active Comparator): This group will receive a pamphlet from the American Institute for Cancer Research (AICR) on dietary prevention and the results of their own breath test, Veggie Meter score and anthropometric measures.
  Interventions: Behavioral: Eating Plan 1
- Eating Plan 2 (Experimental): This group will receive the MyBestGI App and User Manual that encourages limiting four food groups: three or less foods each day made with refined flour, no more than 8% of calories from added sugars, no processed meats and less than 18 oz./week red meat. They will also receive the results of their own breath test, Veggie Meter score and anthropometric measures.
  Interventions: Behavioral: Eating Plan 2
- Eating Plan 3 (Experimental): This group will receive a version of the MyBestGI App and User Manual that encourages meeting 11 food group goals: four food groups to limit and seven food groups to encourage. The 7 groups to encourage are: 3-4 cups/day fruits and vegetables, at least one dark orange or dark green vegetable daily, daily allium and culinary herbs, 3-6 oz./day whole grains, 6-8 oz./week foods high in omega-3 fatty acids, 8-10 tsp./day olive oil or the equivalent from other foods high in monounsaturated fats and at least ½ cup/day of legumes or 1 TB/day nut butter. Some of the goals are personalized based on calculated energy needs. They will also receive the results of their own breath test, Veggie Meter score and anthropometric measures.
  Interventions: Behavioral: Eating Plan 3

INTERVENTIONS:
Behavioral: Eating Plan 1 — The goal is to follow a preventive style of eating that is thought to lower the risk of colorectal cancers.
  Arms: Eating Plan 1
Behavioral: Eating Plan 2 — The goal is to follow a preventive style of eating that is thought to lower the risk of colorectal cancers.
  Arms: Eating Plan 2
Behavioral: Eating Plan 3 — The goal is to follow a preventive style of eating that is thought to lower the risk of colorectal cancers.
  Arms: Eating Plan 3

SUMMARY:
The MyBestGI study evaluates three different approaches that could help people eat in healthier ways. The study seeks to enroll 240 overweight and obese persons who have risk factors for colorectal cancers such as a family or personal history of colorectal cancers or adenomatous polyps. The study website is www.MyBestGI.org .

Participants in the study will be asked to follow one of three eating plans, as best they can, for 12 months. Study participants can choose the foods they prefer within healthy food groups. Two of the eating plans involve ten brief telephone support calls and use of a web-based app (MyBestGI App). The study primarily evaluates improvements in eating and any weight change that may result. Secondary goals for the research are to evaluate how changes in eating affect metabolic pathways.

All study participants will receive written materials that encourage making room for preventive foods in your daily eating. All participants also receive the results of their own diet analyses, and results of their own measures at study visits. The measures are the Veggie Meter skin reflectance test, Ketoscan breath test, and body composition measures. Study visits also involve providing a small blood sample from the arm. Study visits are in Ann Arbor at the start of the study, and at 6 and 12 months.

The long-term goal of this research is to provide better options for supporting individuals who seek to achieve and maintain a preventive style of eating.

DETAILED DESCRIPTION:
Despite the large body of research that has identified the impact of diet on cancer risk, little has been done to improve how care is provided to persons who have risk factors for cancer. The MyBestGI study addresses prevention of colorectal cancer, the third most prevalent cancer in the U.S. Colorectal cancer is among the cancers that are most strongly affected by diet and excess adiposity, and incidence is increasing in young people below the age of 40. More efforts need to be directed at providing individuals with the tools needed for achieving and maintaining a preventive style of eating.

Recommendations for cancer prevention from the American Cancer Society and American Institute for Cancer Research include advice to maintain a healthy weight, to consume more plant-based foods, and to limit red meats, processed meats, and foods with added sugar. This study addresses the development of methods that in the future could feasibly be implemented in medical and community settings to assist individuals with risk factors in attaining both the weight management and diet quality goals for prevention of colorectal cancer.

The MyBestGI study seeks to test three dietary interventions in overweight and obese persons who have risk factors for colorectal cancer. Study participants in all groups receive the results of the Veggie Meter, breath ketones using Ketoscan and body composition testing (InBody270) at study visits. A small blood sample from the arm is taken at each visit for research on how eating affects metabolism.

The MyBestGI study will recruit 240 participants who will be randomized to receive to 12 months of: 1) Eating Plan 1, a group that receives written information on cancer preventive diets; 2) Eating Plan 2 that encourages limiting and logging four food groups associated with increased risks, namely foods containing refined flour, added sugars, processed meats, and red meats; or 3) Eating Plan 3 that combines logging of both food groups to limit and preventive food groups to encourage. Eating Plans 2 and 3 will be supported by written educational materials, brief telephone support calls, and the MyBestGI app. The main outcome is to evaluate to what extent these methods improve eating and possibly achieve weight loss over the year of study.

ELIGIBILITY:
Inclusion Criteria

* Persons ages 19 and older
* The subject has been properly informed of the study, they agree to participate, and sign the Informed Consent document(s)
* Measured body mass index of 25-45 kg/m2 at the study eligibility visit months OR waist circumference > 88 cm for women or > 102 cm for men.
* Reasonably stable weight in the last two months
* Increased risk of colorectal cancer as defined by: Prior adenomatous polyp or serrated polyp OR prior resected early stage CRC (Stage I-IIIA or T1-3, N0-1, M0) OR a history of CRC in at least one primary relative or in at least two secondary relatives OR a polyp was found with a recommended follow-up colonoscopy in less than 8 years OR A known genetic condition that increases risk of CRC
* Good general health
* Have reasonable control over their own dietary intakes
* Not expecting major lifestyle changes in the next 12 months.
* Not expecting a change in hormonal therapies over the next 12 months
* Have and use a smartphone with web access
* Can be contacted by telephone for support calls
* Read and speak English
* Are able to follow a diet high in fiber-containing foods
* Agree to be randomized to a control condition of usual care versus a dietary intervention involving app use and telephone contacts
* Successfully complete three 24-hour dietary recalls online prior to baseline with plausible dietary intakes
* If taking medications for conditions that are affected by diet (diabetes, high blood pressure) must be willing to continue to follow-up with their personal medical provider as needed to manage those conditions and the medication dosing, which may need to be adjusted due to diet changes.
* Has been properly informed of the study and signed the Informed Consent document

Exclusion Criteria:

* Persons with BMI >45 kg/m2 since very high BMI values could indicate more prevalent health problems.
* On medically prescribed diets or other medical contraindications to dietary modification
* Are within 12 months of bariatric surgery
* Pregnant or lactating women or women contemplating pregnancy for the duration of the protocol
* Taking anti-coagulants that interfere with ability to obtain a blood sample
* Has a history of cytotoxic treatment (radiation, chemotherapy) for any type cancer within the last 12 months, except for basal cell or squamous cell tumors of the skin that have been surgically excised and required no further treatment
* Have cancer at the present time
* Dietary intakes with substantial nutrient deficiencies that would require extensive counseling to correct, such as obtaining a large portion of calories from alcohol
* Unable to make their own daily food choices
* Showing evidence of lack of reliability or non-adherence to study procedures (for example, missing an eligibility screening or baseline enrollment appointment more than twice; unable to recall the previous day's diet)
* Reported dietary intakes reported that are not plausible or highly unusual as reported on the ASA24 (for example: <500 or >3500 kcal/day for women and <800 or >4200 kcal/day for men; or reporting too few foods eaten)
* Has an infectious disease at the present time (such as HIV or hepatitis C).
* Unable to read, write, or speak English
* Unable to give informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Preventive Food Score | Change over 12 months
  a score of 10 dietary components (0-10, with 10 being the most optimal score)
Weight Loss | Change over 12 months
  change in weight from baseline (in pounds)

OTHER OUTCOMES:
Breath Ketone Concentration | Change over 12 months
  Ketoscan measure
Skin Carotenoids | Change over 12 months
  Veggie Meter reading

CONTACTS AND LOCATIONS:
Overall Officials: Zora Djuric, PhD, Study Chair — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
This clinical trial will collect data and blood samples from people enrolled in the trial. The study team is open to sharing de-identified data for collaborative work if the scope of the project falls within what was stated in the consent document used for the study. De-identified, aggregate data will also be available upon request for preparation of review articles and meta-analyses. If biosamples are available for sharing after completion of study measures, all sharing and transfer of human data and biospecimens will occur in accordance with sound scientific and ethical principles and shall comply with all applicable laws, regulations, and the policies of the National Institutes of Health and the University of the Michigan.
Supporting Information: Study Protocol, ICF
Time Frame: The primary endpoint data is anticipated to be available by the end of 2026.
Access Criteria: The proposed research use must fall within what is allowed by the consent form.

DOCUMENTS (1):
  • Informed Consent Form (2025-05-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT05396846/ICF_000.pdf